CLINICAL TRIAL: NCT02190253
Title: Seroprevalence of Hepatitis E in The Organ Transplant Subjects
Brief Title: Seroprevalence of Hepatitis E in People With an Organ Transplant
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Georgetown University (Other); University of Pennsylvania (Other); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914148; 14-DK-N148
Record Dates: First submitted 2014-07-12; First posted 2014-07-15 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-05-07

CONDITIONS: Hepatitis E
Keywords: Renal Threshold; Liver Transplant; Transplantation; Hepatitis E; Natural History
MeSH Terms: conditions — Hepatitis E

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Organ transplant recipients: Recipients of either liver, kidney, liver and kidney, and small bowel transplants
- Waitlist patients: Patients on waitlist for liver, kidney or intestinal transplantation

SUMMARY:
Background:

- The hepatitis E virus causes an acute hepatitis that usually goes away by itself. Researchers in France studied people who received a liver or kidney transplant. They found that hepatitis E may not go away by itself in these people. It becomes chronic. This can cause serious liver disease. More than half the people who had organ transplant who had hepatitis E seemed to get a chronic infection.

Researchers want to find out if hepatitis E happens this often in patients who have liver, kidney, or small bowel transplants in the United States. If it does, they want to know why. They want to know if chronic hepatitis E will become an important medical problem. This research might help improve care for people who have a transplant. It also might help researchers prevent the spread of hepatitis E.

Objective:

- To see how many patients who have received or are waiting for certain transplants have antibodies to hepatitis E virus.

Eligibility:

- Adults over age 18 who have had a liver, kidney, liver and kidney, or small bowel transplant, or are on a waiting list for one.

Design:

* Participants will be enrolled from 3 transplant centers.
* Participants will complete a questionnaire. They will be asked about possible risk factors for hepatitis E exposure.
* Participants will have a blood sample drawn through a needle placed in a vein.

DETAILED DESCRIPTION:
Hepatitis E virus infection commonly presents as an acute self-limiting hepatitis in the developing world. However there have been reports that chronic hepatitis E may develop in immunocompromised subjects such as renal and liver transplant recipients. Progression to cirrhosis has also been reported in patients with chronic hepatitis E infection. We hypothesize that immunosuppression post-organ transplantation predisposes individuals to increased susceptibility to hepatitis E infection. Therefore, in this study, we wish to determine the seroprevalence of antibody to hepatitis E IgG in organ transplant recipients (an immunosuppressed population) and compare it to patients who are on organ transplant waitlist (not immunosuppressed). We plan to study samples and date from 300 organ transplant recipients and 300 patients on waitlist for liver, kidney or intestinal transplantation and control for age, gender, organ and transplant center. Three transplant centers (2 in the mid-Atlantic area and one in the Mid-West) will each enroll 100 cases and controls. A minimum of 50 cases at each site will be liver transplant recipients. Cases will be stratified based on number of years post transplant one, two or greater than or equal to three years. Consecutive patients who are eligible and agree to participate in the study will be enrolled. A brief questionnaire to assess risk factors for acquisition of hepatitis E will be administered and 8mls of blood will be drawn in a serum separator tube for anti HEV IgG, anti HEV IgM and HEV RNA testing analysis at the NIH. Subjects who are confirmed to have acute or chronic HEV infection will be managed according to standard of care at each respective transplant centers.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

Inclusion criteria for post-transplant subjects

* Age greater than or equal to 18 years, male or female
* Recipients of either liver, kidney, liver and kidney, and small bowel transplants
* Survival for a minimum of 1 year post-transplant
* Willingness to provide written, informed consent

Exclusion criteria for post-transplant subjects:

* Current or previous treatment within the last year with peg-interferon and or ribavirin.
* Known history of hepatitis E infection.

Inclusion criteria for waitlist subjects:

* Age greater than or equal to 18 years, male or female
* Subjects on the waitlist for first liver, kidney, liver and kidney or small bowel transplant
* Willingness to provide written, informed consent

Exclusion criteria for waitlist subjects:

* Current or previous treatment within the last year with peg-interferon and or ribavirin.
* Current immunosuppression
* Known history of hepatitis E infection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary referral center with liver transplant program
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2014-07-12 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

PRIMARY OUTCOMES:
Seroprevalence of anti-HEV | Baseline
  Seroprevalence of antibody to hepatitis E IgG

CONTACTS AND LOCATIONS:
Overall Officials: Marc G Ghany, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (3):
- United States (3):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Pischke S, Wedemeyer H. Chronic hepatitis E in liver transplant recipients: a significant clinical problem? Minerva Gastroenterol Dietol. 2010 Jun;56(2):121-8. PMID 20485250
- [Background] Gerolami R, Moal V, Picard C, Colson P. Hepatitis E virus as an emerging cause of chronic liver disease in organ transplant recipients. J Hepatol. 2009 Mar;50(3):622-4. doi: 10.1016/j.jhep.2008.12.008. Epub 2008 Dec 25. No abstract available. PMID 19157619
- [Background] Haagsma EB, Niesters HG, van den Berg AP, Riezebos-Brilman A, Porte RJ, Vennema H, Reimerink JH, Koopmans MP. Prevalence of hepatitis E virus infection in liver transplant recipients. Liver Transpl. 2009 Oct;15(10):1225-8. doi: 10.1002/lt.21819. PMID 19790147